CLINICAL TRIAL: NCT00221195
Title: A Prospective, Randomized, Cross-over Study of an Activated Prothrombin Complex Concentrate for Secondary Prophylaxis in Patients With Hemophilia A and Inhibitors
Brief Title: Efficacy Study of Activated Prothrombin Complex for Prevention of Bleeds in Hemophilia A With Inhibitors
Acronym: ProFEIBA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PRO-FEIBA Study
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Hemophilia A With Inhibitors
MeSH Terms: interventions — anti-inhibitor coagulant complex

ARMS (2):
- On-demand first (Other): Patients receive 6 months of on-demand therapy with study drug followed by 6 months of prophylaxis therapy with study drug
  Interventions: Drug: activated prothrombin complex concentrate (FEIBA)
- Prophylaxis first (Other): Patients receive 6 months of prophylaxis therapy with study drug followed by 6 months on-demand therapy with study drug
  Interventions: Drug: activated prothrombin complex concentrate (FEIBA)

INTERVENTIONS:
Drug: activated prothrombin complex concentrate (FEIBA) — FEIBA for prophylaxis therapy dosed at 85 U/Kg +/- 15% on three non-consecutive days each week for 6 months
  FEIBA for on-demand therapy dosed at 85 U/Kg +/- 15% for bleeding episodes for 6 months

SUMMARY:
The objective of this study is to assess whether prophylactic therapy with an activated prothrombin complex concentrate (FEIBA)will result in a significant reduction in the number of bleeds in patients with hemophilia and persistent high responding inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* hemophilia A, any severity, with documented history of high-titer inhibitor (>5BU); current use of bypassing agents (PCCs, aPCCs or rFVIIa) for treatment of bleeds; >/= 6 bleeds requiring bypassing therapy in the previous 6 months

Exclusion Criteria:

* concomitant immune tolerance therapy; clinically symptomatic liver disease, platelet count less than 100,000

Min Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2003-06; Primary Completion 2009-12 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy A Leissinger, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane University School of Medicine, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Gringeri A, Leissinger C, Cortesi PA, Jo H, Fusco F, Riva S, Antmen B, Berntorp E, Biasoli C, Carpenter S, Kavakli K, Morfini M, Negrier C, Rocino A, Schramm W, Windyga J, Zulfikar B, Mantovani LG. Health-related quality of life in patients with haemophilia and inhibitors on prophylaxis with anti-inhibitor complex concentrate: results from the Pro-FEIBA study. Haemophilia. 2013 Sep;19(5):736-43. doi: 10.1111/hae.12178. Epub 2013 Jun 4. PMID 23731246
- [Derived] Leissinger C, Gringeri A, Antmen B, Berntorp E, Biasoli C, Carpenter S, Cortesi P, Jo H, Kavakli K, Lassila R, Morfini M, Negrier C, Rocino A, Schramm W, Serban M, Uscatescu MV, Windyga J, Zulfikar B, Mantovani L. Anti-inhibitor coagulant complex prophylaxis in hemophilia with inhibitors. N Engl J Med. 2011 Nov 3;365(18):1684-92. doi: 10.1056/NEJMoa1104435. PMID 22047559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 16 hemophilia treatment centers in Europe and the United States.
Pre-assignment Details: Patients were randomized to one of two 6 month treatment periods. Following the initial treatment period each subject had a 3 month wash-out period during which time they used on-demand therapy to treat bleeding. Following the 3 month wash-out period each patient was crossed-over to the other 6 month treatment period.
Period: Therapy 1 (Months 1-6)
Arm/Group | On-demand First | Prophylaxis First
Started | 17 | 17
Completed | 14 | 15
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Washout Period (Months 7-9)
Arm/Group | On-demand First | Prophylaxis First
Started | 14 | 15
Completed | 14 | 14
Not Completed | 0 | 1
Not completed — Death | 0 | 1
Period: Therapy 2 (Months 10-15)
Arm/Group | On-demand First | Prophylaxis First
Started | 14 | 14
Completed | 12 | 14
Not Completed | 2 | 0
Not completed — Death | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | On-demand First | Prophylaxis First | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 7 | 11
  Between 18 and 65 years | 13 | 9 | 22
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (13.4) | 24.9 (20.6) | 27.1 (17.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 17 | 34
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
  Europe | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Bleeds During 6 Month Treatment Period
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: bleeds
Groups:
- Bleeds During the On-demand Period: During the on-demand period, bleeding was treated with AICC at a target dose of 85 U per kilogram of body weight (±15%) (range, 72 to 98). For bleeding episodes that did not respond to the specified therapy, alternative treatment, including additional doses of AICC, rFVIIa, or factor VIII, was allowed at the discretion of the treating physician.
  Final analysis only included those who completed per protocol, only 26 subjects completed the study.
- Bleeds During the Prophylaxis Period: During the prophylaxis period, AICC was administered at a target dose of 85 U per kilogram (±15%) (range, 72 to 98) on 3 nonconsecutive days weekly. Bleeding episodes during the prophylaxis period were treated with AICC at a target dose of 85 U per kilogram of body weight (±15%) (range, 72 to 98). For bleeding episodes that did not respond to the specified therapy, alternative treatment, including additional doses of AICC, rFVIIa, or factor VIII, was allowed at the discretion of the treating physician.
  Final analysis only included those who completed per protocol, only 26 subjects completed the study.
Arm/Group | Bleeds During the On-demand Period | Bleeds During the Prophylaxis Period
Number analyzed (Participants) | 26 | 26
bleeds | 13.1 (7.1) | 5.0 (5.0)
Statistical Analysis 1: Comparison: Bleeds During the On-demand Period vs Bleeds During the Prophylaxis Period; The Wilcoxin signed-rank test was used to compare the frequency of bleeds between the prophylaxis and on-demand periods; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of consent to the end of the study, which totaled 15 months.
Groups:
- On-demand Period: During the on-demand period, bleeding was treated with AICC at a target dose of 85 U per kilogram of body weight (±15%) (range, 72 to 98). For bleeding episodes that did not respond to the specified therapy, alternative treatment, including additional doses of AICC, rFVIIa, or factor VIII, was allowed at the discretion of the treating physician.
  There were 3 subjects that never received on-demand therapy, therefore 31 subjects were assessed for AEs during this period.
- Prophylaxis Period: During the prophylaxis period, AICC was administered at a target dose of 85 U per kilogram (±15%) (range, 72 to 98) on 3 nonconsecutive days weekly. Bleeding episodes during the prophylaxis period were treated with AICC at a target dose of 85 U per kilogram of body weight (±15%) (range, 72 to 98). For bleeding episodes that did not respond to the specified therapy, alternative treatment, including additional doses of AICC, rFVIIa, or factor VIII, was allowed at the discretion of the treating physician.
  There were 3 subjects that never received prophylaxis therapy, therefore 31 subjects were assessed for AEs during this period.
- Washout Period: Bleeding episodes during the washout period were treated with AICC at a target dose of 85 U per kilogram of body weight (±15%) (range, 72 to 98). For bleeding episodes that did not respond to the specified therapy, alternative treatment, including additional doses of AICC, rFVIIa, or factor VIII, was allowed at the discretion of the treating physician.
  There were 5 subjects that never entered the washout period, therefore 31 subjects were assessed for AEs during this period.
Arm/Group | On-demand Period | Prophylaxis Period | Washout Period
Serious Adverse Events (participants affected / at risk) | 3/31 | 4/31 | 4/29
Other Adverse Events (participants affected / at risk) | 16/31 | 17/31 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | On-demand Period (N=31) | Prophylaxis Period (N=31) | Washout Period (N=29)
Chest Pain (Cardiac disorders) | 0 | 1 | 0
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Drug hypersensitivity (Product Issues) | 0 | 1 | 0
Phlebitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Hospitalization (Endocrine disorders) | 1 | 0 | 0
Surgical Procedure (Surgical and medical procedures) | 1 | 0 | 0
Catheter-site Hemorrhage (Blood and lymphatic system disorders) | 1 | 1 | 0
Catheter-site Infection (Infections and infestations) | 1 | 2 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Cerebral Hemorrhage (Vascular disorders) | 0 | 0 | 1
Subdural Hematoma (Vascular disorders) | 0 | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle Hemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | On-demand Period (N=31) | Prophylaxis Period (N=31) | Washout Period (N=29)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Headache (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Pyrexia (General disorders) | 2 | 6 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 2 | 0 | 0
Ecchymosis (Blood and lymphatic system disorders) | 2 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 2
Influenza (Infections and infestations) | 1 | 1 | 4
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Upper Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1
Poor Venous Access (Surgical and medical procedures) | 0 | 1 | 0
Catheter-site Hemorrhage (Blood and lymphatic system disorders) | 1 | 2 | 0
Catheter-site Infection (Infections and infestations) | 1 | 2 | 0
Staphylococcal Infection (Infections and infestations) | 1 | 0 | 0
Tongue Hemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
One limitation was the relatively short duration; in addition, due to the small number of children enrolled, it is not possible to draw conclusions regarding the relationship of age and the benefits of prophylaxis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less